CLINICAL TRIAL: NCT00355290
Title: Changes in Oral Vitamin K Intake for Optimization of Chronic Oral Anticoagulation: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCPA2006.01
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Blood Coagulation Disorders
Keywords: Chronic Oral Anticoagulation
MeSH Terms: conditions — Blood Coagulation Disorders

INTERVENTIONS:
Behavioral: Changes on Oral Vitamin K Intake

SUMMARY:
The primary hypothesis of this trial is that changes in oral vitamin K intake, based on simple food registries, may be superior to conventional changes in doses of medications in order to stabilize chronic oral anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any clinical indication for chronic oral anticoagulation with one INR level out of target, without a clear clinical cause for INR instability (unplanned changes in coumadin medications, other pharmacological interactions, clinical illnesses and laboratory errors).

Exclusion Criteria:

* Clinical evidence of bleeding or thrombosis.
* INR > 4 or INR < 1,5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2006-08; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients on target International Normalized Ratio (prothrombin time) on day 90th after randomization
Stabilization of International Normalized Ratio (prothrombin time) during follow-up (90 days after randomization)

CONTACTS AND LOCATIONS:
Overall Officials: Luis E Rohde, MD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] de Assis MC, Rabelo ER, Avila CW, Polanczyk CA, Rohde LE. Improved oral anticoagulation after a dietary vitamin k-guided strategy: a randomized controlled trial. Circulation. 2009 Sep 22;120(12):1115-22, 3 p following 1122. doi: 10.1161/CIRCULATIONAHA.109.849208. Epub 2009 Sep 8. PMID 19738137